CLINICAL TRIAL: NCT05636397
Title: A Phase I, Safety and Pharmacokinetics/pharmacodynamics Study of Oral L-CIT Supplementation in Preterm Infants with BPD±PH and NEC
Brief Title: Safety and PK-PD Study of Oral L-CIT in Preterm Infants with BPD±PH and NEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Estelle Gauda, Head, Division of Neonatology, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000077413
Record Dates: First submitted 2022-10-26; First posted 2022-12-05 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: BPD - Bronchopulmonary Dysplasia; Pulmonary Hypertension; NEC
Keywords: BPD±PH; surgical NEC; L-Citrulline; Pharmacokinetic profile; Pharmacodynamic profile; Preterm neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: This is a prospective dose-escalation study.
  Arm 1: BPD-PH Total of 12-24 infants; 6-12 at each dose level. (300 or 500 mg/kg/day divided q6 hours)
  Arm 2: sNEC A total of 18-36 infants with Stage III NEC; 6-12 at each dose level. (75, 150 or 225 mg/kg/day divided q6 hours)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPD±PH (Experimental): Arm 1: BPD±PH
  Total of 12-24 infants; 6-12 at each dose level of oral dosage form of L-Citrulline. (300 or 500 mg/kg/day divided q6 hours).
  Dose Level 1 = 300 mg/kg/day Dose Level 2 = 500 mg/kg/day
  Interventions: Dietary Supplement: L-Citrulline
- Surgical NEC (Experimental): Arm 2: sNEC
  A total of 18-36 infants with Stage III NEC; 6-12 at each dose level of oral dosage form of L-Citrulline. (75, 150 or 225 mg/kg/day divided q6 hours)
  Dose Level 1 = 75 mg/kg/day Dose Level 2 = 150 mg/kg/day Dose Level 3 = 225 mg/kg/day
  Interventions: Dietary Supplement: L-Citrulline

INTERVENTIONS:
Dietary Supplement: L-Citrulline — Citrulline is a nonessential amino acid made in the small intestine, occurs naturally in the body, and is believed to help reduce inflammation.L-CIT is a part of the urea cycle, produced as a by-product along with nitric oxide (NO).

SUMMARY:
The purpose of this study is to evaluate the safety and explore the PK/PD of L-CIT supplementation in preterm infants to prevent the development of inflammatory pathways initiated by low levels of plasma CIT, specifically in preterm infants with post surgical NEC and BPD±PH.

DETAILED DESCRIPTION:
Preterm infants are born with underdeveloped organs and immune systems, placing them at great risk for morbidity. They are more susceptible to inflammatory injury, particularly from conditions of prematurity mediated by inflammatory pathways such as bronchopulmonary dysplasia (BPD) and necrotizing enterocolitis (NEC).

L-CIT, an amino acid, is the first intermediate in the urea cycle as well as a precursor to arginine and nitric oxide (NO), which promotes blood flow. It is made in the intestine and has been shown to exert vasoprotective and anti-inflammatory effects. BPD-PH and NEC are two specific inflammatory diseases of prematurity involving CIT, arginine or NO deficiencies.

Evaluation of the safety and PK/PD of L-CIT supplementation for diseases involving CIT, arginine or NO deficiencies in preterm infants is important. Therefore, in this trial the investigator would like to evaluate the safety and pharmacokinetics/pharmacodynamics (PD) of L-CIT supplementation in preterm infants post surgical NEC and BPD-PH.

ELIGIBILITY:
Arm 1: BPD±PH:

Inclusion Criteria:

* Born ≤ 30 weeks at birth
* Post-menstrual age (PMA) ≥ 34 weeks
* Echocardiographic evidence of PH for infants with BPD+PH
* On invasive or non-invasive ventilation with RSS >2.0 for >12hours/day for at least 48 hours
* Informed written consent (parents/substitute decision maker)

Exclusion Criteria:

* Congenital Heart Disease [Exceptions: small atrial septal defect (ASD), small ventricular septal defect (VSD), small patent ductus arteriosus (PDA)]
* Infants with pulmonary vein stenosis
* Concurrent sepsis with hemodynamic instability
* Infants considered likely to die within next 7 days
* Any other condition that, in the opinion of the investigator, may adversely affect the infant's ability to complete the study or its measures or pose significant risk to the infant.

Arm 2: surgical NEC

Inclusion Criteria

* Born ≤ 30 weeks at birth
* Recovering from Stage IIIb NEC as per modified Bell's staging (pneumoperitoneum requiring surgery)
* Tolerating 30 ml/kg/day of enteral feeds
* On invasive or non-invasive ventilation (NIPPV/nCPAP) with RSS >2.0 for > 12hours/day for at least 48 hours, 10-14 days post surgery
* Informed written consent (parents/substitute decision maker)
* Considered medically stable by clinical team

Exclusion Criteria:

* Congenital heart disease (except small ASD, small VSD and non hsPDA)
* Pulmonary vein stenosis
* Concurrent sepsis with hemodynamic instability
* Likely to die within next 7 days
* Other condition significantly affecting pulmonary function independent of prematurity or NEC

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety of oral L-Citrulline administration | 5 years
  The number of patients with adverse events (AE) as a measure of safety and tolerability

SECONDARY OUTCOMES:
Association of blood pressure as one of the PD outcomes with maximum L-CIT concentration (Cmax) | 5 years
  Blood pressure of the study participants will be associated with PK measures of L-CIT exposure i.e. Cmax using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Association of stoma or nasogastric output as one of the PD outcomes with maximum L-CIT concentration (Cmax) | 5 years
  Stoma or nasogastric output of the study participants will be associated with PK measures of L-CIT exposure i.e. Cmax using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Association of stool output as one of the PD outcomes with maximum L-CIT concentration (Cmax) | 5 years
  Stool output from the study participants will be associated with PK measures of L-CIT exposure i.e. Cmax using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Association of blood pressure with the area under the concentration time curve (AUC) for L-CIT | 5 years
  Blood pressure of the study participants will be associated with PK measures of L-CIT exposure i.e. Area under Concentration time curve (AUC) using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen.
Association of stoma or nasogastric output with the area under the concentration time curve (AUC) for L-CIT | 5 years
  Stoma or nasogastric output of the study participants will be associated with PK measures of L-CIT exposure i.e. Area under Concentration time curve (AUC) using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen.
Association of stool output with the area under the concentration time curve (AUC) for L-CIT | 5 years
  Stool output from the study participants will be associated with PK measures of L-CIT exposure i.e. Area under Concentration time curve (AUC) using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen.
Association of blood pressure with minimum L-CIT concentration (Cmin) | 5 years
  Blood pressure of study participants will be associated with PK measures of L-CIT exposure i.e. Cmin using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Association of stoma or nasogastric output with minimum L-CIT concentration (Cmin) | 5 years
  Stoma or nasogastric output from study participants will be associated with PK measures of L-CIT exposure i.e. Cmin using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Association of stool output with minimum L-CIT concentration (Cmin) | 5 years
  Stool output from study participants will be associated with PK measures of L-CIT exposure i.e. Cmin using univariate correlation approaches. The investigator will then attempt to construct a PK/PD model to link PK and PD measures found to be of significance during the univariate screen. Future larger studies will then be used to examine these relationships with adequately powered studies.
Correlation between CIT and arginine levels | 5 years
  Correlation between changes in CIT and arginine levels with nitrite/nitrate levels
Biomarkers of inflammation | 5 years
  The levels of IL-1β, IL-6, IL-8, IL-10, TNFα will be measured in tracheal aspirates and blood plasma. The aggregated levels fo these cytokines will reflect the inflammatory status of the study participant.
Oxidative stress | 5 years
  Oxidative stress (measured in tracheal aspirates and blood)
Respiratory Score (RSS) | 5 years
  The respiratory severity score (RSS) is a simplified severity score consisting of the mean airway pressure (MAP) multiplied by the fraction of inspired oxygen (FiO2). This score ranges from 0 to 12, with a higher score indicating more severe lung disease.
Desaturation index | 5 years
  The oxygen desaturation index (ODI) is commonly used to evaluate the severity of nocturnal hypoxemia. The ODI is defined as the number of episodes of oxygen desaturation per hour of sleep with desaturation events of >=10sec/ sampled hour.
Changes in Blood Pressure | 5 years
  Changes in diastolic and systolic blood pressure prior to and during CIT treatment.
Stoma, nasogastric or stool output | 5 years
  Volume of stoma, nasogastric or stool output prior to and during CIT treatment
Ventilation | 5 years
  Days on mechanical ventilation, non-invasive ventilation, and supplementary oxygen
BPD severity | 5 years
  Moderate to severe BPD based on the different mode of ventilatory support needed at 36 wks PMA.
  No BPD = off all oxygen and positive pressure support Moderate BPD = low flow oxygen only Severe BPD= positive pressure support (high flow, CPAP, NIPPV, or ETT)
BPD | 5 years
  number of days of survival free of BPD
Pre-discharge mortality | 5 years
  Number of study participants who died during NICU admission.
Postnatal steroid Use | 5 years
  Number of days study participants received postnatal steroids during their NICU stay.
Bayley's scale for infant development | 5 years
  Bayley Scales of Infant and Toddler Development is an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood. BSID is the commonly used abbreviation for Bayley Scales of Infant and Toddler Development. Bayley-III includes a motor score, and fine and gross motor subtest scores. The standardized mean motor score is 100 (SD 15), with scores lower than 85 indicating mild impairment, and lower than 70 indicating moderate or severe impairment.In this particular trial, the investigator would be looking at the correlation between the inflammatory markers (IL-1β, IL-6, IL-8, IL-10, TNFα) and Neurodevelopmental outcomes from Bayley's scale during 18-24M follow up visit in babies received L-Citrulline during their NICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Gauda, MD, Principal Investigator — Division Head, Division of Neonatology
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.